CLINICAL TRIAL: NCT04138667
Title: Investigation and Comparison of Lymphedema Outcome Measurements Validated in Turkish for Assessment of Breast Cancer Related Lymphedema
Brief Title: Responsiveness of Outcome Scales in Breast Cancer Related Lymphedema
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 09.2019.865
Record Dates: First submitted 2019-10-19; First posted 2019-10-24 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Lymphedema of Upper Arm
Keywords: breast cancer related lymphedema; lymphedema; outcome measurement; responsiveness
MeSH Terms: conditions — Breast Cancer Lymphedema; Lymphedema

STUDY DESIGN:
Intervention Model Description: Patients with breast cancer related lymphedema who will undergo complex decongestive phase 1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with post-mastectomy lymphedema (Experimental): Patients with breast cancer related lymphedema who will undergo complex decongestive therapy
  Interventions: Other: complex decongestive therapy

INTERVENTIONS:
Other: complex decongestive therapy — Complex decongestive therapy-phase 1 program consist of meticulous skin and nail care, manuel lymphatic drainage, compression bandages, and remedial exercises. All patients will receive manual lymphatic drainage for three times a week (Monday-Wednesday-Friday) during 4 weeks, 50 minutes a day (a total of 12 sessions) by a trained lymphatic massage therapist.

SUMMARY:
The aim of this study is to investigate and compare responsiveness of current lymphedema assessment scales validated in Turkish.

DETAILED DESCRIPTION:
Lymphedema is defined as the excessive and persistent accumulation of fluid, extracellular proteins, and fat in tissue spaces, caused by inefficiency of the lymphatic drainage system. It is a chronic, progressive condition. Several researchers have investigated the influence on health-related quality of life in upper limb lymphedema after breast cancer treatment using patient reported outcome instruments. Responsiveness of only one of the lymphedema assessment scale, ''Lymphedema Quality of Life Inventory'', has been investigated. Responsiveness of lymphedema assessment scales validated in Turkish has not been examined in detail, thereby limiting their use in clinical trials. Therefore, the aim of this study is to investigate and compare responsiveness of current lymphedema assessment scales validated in Turkish. Patients with breast cancer related lymphedema with International Society of Lymphology-ISL lymphedema stage 2,3 will be included in the study and will receive complex decongestive therapy phase I including meticulous skin and nail care, manuel lymphatic drainage, compression bandages, and remedial exercises. All patients will receive manual lymphatic drainage for three times a week (Monday-Wednesday-Friday) during 4 weeks, 50 minutes a day (a total of 12 sessions) by a trained lymphatic massage therapist. Limb volume will be calculated based on truncated cone method from circumference measurements. Patients will complete Lymphedema Life Impact Scale (LLIS), Patient Benefit Index-Lymphedema(PBI), Lymphedema functioning, disability and health questionnaire(Lymph-ICF), European Organization for Research and Treatment of Cancer Quality of Life Breast Cancer (EORTC-QLQ-30) and Short Form 36 (SF-36) before and after treatment. Changes in limb volumes will be compared in changes in scales after treatment. Responsiveness of the subscales will be will be determined by calculating the effect size (change in all patients), standardized mean response (effect size in a group with improvement), and Guyatt's Responsiveness Index.

ELIGIBILITY:
Inclusion Criteria:

-Patients with unilateral postmastectomy lymphedema with a International Society of Lymphology-ISL) stage 2 and 3

Exclusion Criteria:

* Bilateral lymphedema
* The patients who had known systemic edematogenic conditions (e.g., cardiac/hepatic/renal failure, terminal cancer, on chemotherapy), and/or with cancer recurrence
* Patients with contraindications for application of complex decongestive therapy (active cutaneous infection, deep vein thrombosis, cardiac edema, and peripheral artery disease)

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-10-19 (Actual); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-05-30 (Estimated)

PRIMARY OUTCOMES:
Limb volume measurement | before treatment (T0)
  Limb volume will be calculated based on truncated cone method from circumference measurements
Limb volume measurement | after treatment (T1) (through completion of four weeks of complex decongestive therapy phase 1)
  Limb volume will be calculated based on truncated cone method from circumference measurements

SECONDARY OUTCOMES:
Lymphedema Quality of Life Questionnaire-Arm (LYMQOL) | before treatment (T0)
  The LYMQOL-Arm has been developed to assess the impact of lymphedema of the arms on the QoL of the patients. It consists of four domains with 28 items. These domains are symptoms, appearance, function, and mood. The answers were evaluated on a four-point Likert scale (1= not at all 2= a little, 3= quite a bit, 4= a lot). Each item received a score between 1 and 4, with higher scores indicating a worse QoL.
Lymphedema Quality of Life Questionnaire-Arm | after treatment (T1) (through completion of four weeks of complex decongestive therapy phase 1)
  The LYMQOL-Arm has been developed to assess the impact of lymphedema of the arms on the QoL of the patients. It consists of four domains with 28 items. These domains are symptoms, appearance, function, and mood. The answers were evaluated on a four-point Likert scale (1= not at all 2= a little, 3= quite a bit, 4= a lot). Each item received a score between 1 and 4, with higher scores indicating a worse QoL.
Lymphedema Life Impact Scale (LLIS) | before treatment (T0)
  The LLIS is an 18-item measure of physical, psychosocial, and functional impairments caused by lymphedema.
Lymphedema Life Impact Scale (LLIS) | after treatment (T1) (through completion of four weeks of complex decongestive therapy phase 1)
  The LLIS is an 18-item measure of physical, psychosocial, and functional impairments caused by lymphedema.
Patient Benefit Index-Lymphedema(PBI) | before treatment (T0)
  The Patient Benefit Index (PBI) methodology allows for a more direct measurement of patient-relevant treatment.benefit. In the first part the Patient Needs Questionnaire (PNQ)patients rate the importance of a list of patient relevant treatment goals on a five-step scale from "not at all" to "very". In the second part the Patient Benefit Questionnaire (PBQ) patients rate to what extent the treatment goals have been achieved on the same five-step scale. Alternatively, they can choose "does not apply to me" for each treatment goal in both questionnaires. Thus, the patient directly evaluates treatment benefit instead of rating her/his current HRQoL before and after treatment. A PBI weighted global score ranging from 0 (no benefit) to 4 (maximum benefit) is computed for each patient. The weighting algorithm8 ensures that the achievement of important treatment goals will have higher impact on the global score than the achievement of less important goals.
Patient Benefit Index-Lymphedema(PBI) | after treatment (T1) (through completion of four weeks of complex decongestive therapy phase 1)
  The Patient Benefit Index (PBI) methodology allows for a more direct measurement of patient-relevant treatment.benefit. In the first part the Patient Needs Questionnaire (PNQ) patients rate the importance of a list of patient relevant treatment goals on a five-step scale from "not at all" to "very". In the second part the Patient Benefit Questionnaire (PBQ) patients rate to what extent the treatment goals have been achieved on the same five-step scale. Alternatively, they can choose "does not apply to me" for each treatment goal in both questionnaires. Thus, the patient directly evaluates treatment benefit instead of rating her/his current HRQoL before and after treatment. A PBI weighted global score ranging from 0 (no benefit) to 4 (maximum benefit) is computed for each patient. The weighting algorithm8 ensures that the achievement of important treatment goals will have higher impact on the global score than the achievement of less important goals.
Lymphoedema functioning, disability and health questionnaire(Lymph-ICF) | before treatment (T0)
  The Lymph-ICF questionnaire is composed of 29 questions. Each question is answered using a visual analog scale (VAS) ranging from 0 to 100 mm. The anchors for the impairments in function (e.g. "Does your arm hurt?") are "not at all" and "very much," and those for the activity limitations and participation restrictions (e.g. "Are you able to carry heavy weights?") are "very well" and "not at all." The Lymph-ICF has 5 domains: physical function, mental function, household activities, mobility activities, and life and social activities. The total score of the Lymph-ICF is equal to the sum of the scores of the questions divided by the total number of answered questions.
Lymphoedema functioning, disability and health questionnaire(Lymph-ICF) | after treatment (T1) (through completion of four weeks of complex decongestive therapy phase 1)
  The Lymph-ICF questionnaire is composed of 29 questions. Each question is answered using a visual analog scale (VAS) ranging from 0 to 100 mm. The anchors for the impairments in function (e.g. "Does your arm hurt?") are "not at all" and "very much," and those for the activity limitations and participation restrictions (e.g. "Are you able to carry heavy weights?") are "very well" and "not at all." The Lymph-ICF has 5 domains: physical function, mental function, household activities, mobility activities, and life and social activities. The total score of the Lymph-ICF is equal to the sum of the scores of the questions divided by the total number of answered questions.
European Organization for Research and Treatment of Cancer QoL Breast Cancer (EORTC-QLQ-30) | before treatment (T0)
  The EORTC QLQ-C30 questionnaire is a survey conducted to evaluate the quality of life in patients with breast cancer. It consists of 30 questions which assess symptoms that occurred in the previous two weeks. Responses are given on a Likert scale: 1 - not at all, 2 - a little, 3 - quite a bit, 4 - very much. The global health scale consists of two questions asking patients to classify their general health and quality of life in the previous week, by rating it from 1 to 7, in which 1 means poor and 7, excellent. The questionnaires are divided into three scales: global health scale (GHS), functional scale (FS) and symptom scale (SS).
European Organization for Research and Treatment of Cancer QoL Breast Cancer (EORTC-QLQ-30) | after treatment (T1) (through completion of four weeks of complex decongestive therapy phase 1)
  The EORTC QLQ-C30 questionnaire is a survey conducted to evaluate the quality of life in patients with breast cancer. It consists of 30 questions which assess symptoms that occurred in the previous two weeks. Responses are given on a Likert scale: 1 - not at all, 2 - a little, 3 - quite a bit, 4 - very much. The global health scale consists of two questions asking patients to classify their general health and quality of life in the previous week, by rating it from 1 to 7, in which 1 means poor and 7, excellent. The questionnaires are divided into three scales: global health scale (GHS), functional scale (FS) and symptom scale (SS).
Short Form 36 (SF-36) | before treatment (T0)
  The Short Form 36 (SF-36) Health Survey measures overall health. It has eight sections: Physical functioning (10), role limitations due to physical health (4), role limitations due to emotional problems (3), energy/fatigue (4), emotional well-being (5), social functioning (2), pain (2), and general health (5). Each scale is transformed into a 0-100 scale on the assumption that each scale carries equal weight. The lower the score, the more disability.
Short Form 36 (SF-36) | after treatment (T1) (through completion of four weeks of complex decongestive therapy phase 1)
  The Short Form 36 (SF-36) Health Survey measures overall health. It has eight sections: Physical functioning (10), role limitations due to physical health (4), role limitations due to emotional problems (3), energy/fatigue (4), emotional well-being (5), social functioning (2), pain (2), and general health (5). Each scale is transformed into a 0-100 scale on the assumption that each scale carries equal weight. The lower the score, the more disability.

CONTACTS AND LOCATIONS:
Overall Officials: Gulseren Akyuz, Prof, Study Chair — Marmara University
Locations (1):
- Marmara University School of Medicine Department of Physical Medicine and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The investigators don't plan to share individual participant data (IPD) in public.

REFERENCES:
- [Result] Menz HB, Auhl M, Tan JM, Levinger P, Roddy E, Munteanu SE. Comparative Responsiveness of Outcome Measures for the Assessment of Pain and Function in Osteoarthritis of the First Metatarsophalangeal Joint. Arthritis Care Res (Hoboken). 2020 May;72(5):679-684. doi: 10.1002/acr.23883. Epub 2020 Apr 8. PMID 30908853
- [Result] Borman P, Yaman A, Denizli M, Karahan S, Ozdemir O. The reliability and validity of Lymphedema Quality of Life Questionnaire-Arm in Turkish patients with upper limb lymphedema related with breast cancer. Turk J Phys Med Rehabil. 2018 Jul 9;64(3):205-212. doi: 10.5606/tftrd.2018.2843. eCollection 2018 Sep. PMID 31453513
- [Result] Duygu E, Bakar Y, Keser I. An Important Tool in Lymphedema Management: Validation of Turkish Version of the Patient Benefit Index-Lymphedema. Lymphat Res Biol. 2020 Feb;18(1):49-55. doi: 10.1089/lrb.2018.0036. Epub 2019 May 30. PMID 31145018
- [Result] Bakar Y, Tugral A. Translation, reliability, and validation of the Turkish version of the Lymphedema Quality-of-Life tool in Turkish-speaking patients with lower limb Lymphedema. J Vasc Nurs. 2019 Mar;37(1):11-17. doi: 10.1016/j.jvn.2018.11.005. Epub 2019 Jan 31. PMID 30954192
- [Result] Bakar Y, Tugral A, Ozdemir O, Duygu E, Uyeturk U. Translation and Validation of the Turkish Version of Lymphedema Quality of Life Tool (LYMQOL) in Patients with Breast Cancer Related Lymphedema. Eur J Breast Health. 2017 Jul 1;13(3):123-128. doi: 10.5152/ejbh.2017.3522. eCollection 2017 Jul. PMID 28894851
- [Result] Kostanoglu A, Hosbay Z, Tarakci E. Lymphoedema functioning, disability and health questionnaire Turkish version: translation, cross-cultural adaptation and validation. J Phys Ther Sci. 2016 Jun;28(6):1728-32. doi: 10.1589/jpts.28.1728. Epub 2016 Jun 28. PMID 27390404